CLINICAL TRIAL: NCT06787677
Title: The Efficacy and Safety of Sphenopalatine Ganglion Pulsed Radiofrequency Treatment for Chronic Cluster Headache
Brief Title: SPG Pulsed Radiofrequency for Chronic Cluster Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY 2018-027-02-1
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Headache, Cluster
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF group (Experimental)
  Interventions: Procedure: PRF
- Nerve Block Group (Active Comparator)
  Interventions: Procedure: NB

INTERVENTIONS:
Procedure: PRF — After the puncture needle reached the sphenopalatine ganglion (SPG), patients in the PRF group received PRF treatment in automatic mode for 360 s, at a maximum of 42°C, pulse frequency of 2 Hz, and pulse width of 20 ms.
  Arms: PRF group
Procedure: NB — After the puncture needle reached the sphenopalatine ganglion (SPG), patients in the NB group received nerve block with a mixture of 40 mg of triamcinolone and 2 ml of 0.75% bupivacaine with 2 ml of normal saline and 1:100000 epinephrine.
  Arms: Nerve Block Group

SUMMARY:
Cluster headache (CH) is a devastating disorder characterized by ipsilateral headache and associated trigeminal autonomic symptoms, with a yearly prevalence of 0.1%. There is a huge clinically unmet demand for an effective therapeutic method for CH. Previous evidences indicate that pulse radiofrequency (PRF) targeting the sphenopalatine ganglion (SPG) is a safe, minimally invasive, effective treatment for CH. This randomized, controlled trial aimed to establish the safety and efficacy of SPG PRF for patients with chronic CH.

ELIGIBILITY:
Inclusion Criteria:

* Chronic cluster headache;
* At least four attacks per week;
* Minimum age of 18 years;
* Non-response to verapamil and lithium treatment in the past, intolerance, or contraindication to verapamil and lithium, along with non-response, intolerance, or contraindica-tion to topiramate, or gabapentin.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Presence of cardiac pacemaker or other neuromodulatory devices;
* Pyschiatric and cognitive disorders;
* Serious drug habituation or overuse of acute-headache medication;
* History of stroke or intracranial aneurysm, or at risk for serious or acute cardiovascular events;
* Infection at the puncture site;
* Previous history of invasive treatments such as sphenopalatine ganglion radiofrequency thermocoagulation and chemical destruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The mean attack frequency in the last 4 weeks (week 8-12) after procedure | In the last 4 weeks (week 8-12) after procedure
  The overall mean change from baseline in mean weekly attack frequency

SECONDARY OUTCOMES:
Mean attack frequency | From baseline to each 4-week interval through 1 year after procedure
  Mean change in mean attack frequency
50% reduction of mean attack frequency | From baseline to each 4-week interval through 1 year after procedure
  Percentage of patients with a 50% reduction in mean attack frequency
30% reduction of mean attack frequency | From baseline to each 4-week interval through 1 year after procedure
  Percentage of patients with a 30% reduction in mean attack frequency
Patient Global Impression of Improvement | At month 1, month 2, month 3, month 6, and month 12 after procedure
  Percentage of patients reporting a score of 1 (''very much better'') or 2 (''much better'')
Mean attack intensity | From baseline to each 4-week interval through 1 year after procedure
  0-10 on the numeric rating scale, with 0 equating no pain and 10 the worst pain possible
Patient satisfaction scores | At month 1, month 2, month 3, month 6, and month 12 after procedure
  0 point indicates unsatisfied to 10 points indicate very satisfied. The higher the score, the more dissatisfied the patient is.
The incidence of perioperative adverse events | Across 1 year after procedure
  Perioperative adverse events (AEs) including headache, dizziness, nausea, vomiting, facial hematoma, and numbness in the area innervated by the maxillary nerve

CONTACTS AND LOCATIONS:
Locations (1):
- Fang Luo, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.

REFERENCES:
- [Background] Goadsby PJ, Sahai-Srivastava S, Kezirian EJ, Calhoun AH, Matthews DC, McAllister PJ, Costantino PD, Friedman DI, Zuniga JR, Mechtler LL, Popat SR, Rezai AR, Dodick DW. Safety and efficacy of sphenopalatine ganglion stimulation for chronic cluster headache: a double-blind, randomised controlled trial. Lancet Neurol. 2019 Dec;18(12):1081-1090. doi: 10.1016/S1474-4422(19)30322-9. PMID 31701891
- [Result] Schoenen J, Snoer AH, Brandt RB, Fronczek R, Wei DY, Chung CS, Diener HC, Dodick DW, Fontaine D, Goadsby PJ, Matharu MS, May A, McGinley JS, Tepper SJ, Jensen RH, Ferrari MD; IHS Standing Committee for Clinical Trials; IHS cluster headache trial guideline subcommittee. Guidelines of the International Headache Society for Controlled Clinical Trials in Cluster Headache. Cephalalgia. 2022 Dec;42(14):1450-1466. doi: 10.1177/03331024221120266. Epub 2022 Oct 21. PMID 36268950
- [Result] Wilbrink LA, de Coo IF, Doesborg PGG, Mulleners WM, Teernstra OPM, Bartels EC, Burger K, Wille F, van Dongen RTM, Kurt E, Spincemaille GH, Haan J, van Zwet EW, Huygen FJPM, Ferrari MD; ICON study group. Safety and efficacy of occipital nerve stimulation for attack prevention in medically intractable chronic cluster headache (ICON): a randomised, double-blind, multicentre, phase 3, electrical dose-controlled trial. Lancet Neurol. 2021 Jul;20(7):515-525. doi: 10.1016/S1474-4422(21)00101-0. PMID 34146510